CLINICAL TRIAL: NCT03538574
Title: Mindfulness Meditation and Insomnia in Alzheimer Disease Caregivers: Inflammatory and Biological Aging Mechanisms
Brief Title: Mindfulness Meditation and Insomnia in Alzheimer Disease Caregivers
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Irwin, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-001256
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2021-06

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, non-inferiority design
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcome assessor is blind to treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Active Comparator): Cognitive behavioral therapy for insomnia (CBT-I), considered the treatment of choice by the American Academy of Sleep Medicine, combines cognitive therapy, stimulus control, sleep restriction, sleep hygiene, and relaxation to improve sleep outcomes, with demonstrated efficacy in adult and older adult populations
  Interventions: Behavioral: CBT-I
- MAP-I (Experimental): The Mindful Awareness Practices (MAPs) is a validated and curriculum-based meditation similar to Mindfulness Based Stress Reduction, with the exception that MAPs does not include a day-long retreat or yoga and hence takes a more practical and accessible approach that focuses specifically on the practice of mindfulness and its application in everyday life. (http://marc.ucla.edu) MAP for Insomnia (MAP-I) is a modified version of MAPs that incorporates practice prior to bed, use of practice in the bed during night-time awakenings, and daily body scan.
  Interventions: Behavioral: MAP-I

INTERVENTIONS:
Behavioral: CBT-I — CBT-I is a behavioral treatment for insomnia
  Arms: CBT-I
Behavioral: MAP-I — MAP-I is a mindfulness meditation treatment for insomnia
  Arms: MAP-I

SUMMARY:
Treatment of insomnia in caregivers is needed given that 60% of Alzheimer disease caregivers report sleep complaints, and insomnia may add to the burden of AD caregiving and contribute to morbidity and mortality risk. This is the first intervention trial in AD caregivers to target insomnia and also evaluate two mechanisms of chronic disease risk, inflammation and cellular aging

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the non-inferiority of Mindful Awareness Practices for Insomnia (MAP-I ) vs. Cognitive Behavioral Therapy for Insomnia (CBT-I) on outcomes of insomnia, cellular and genomic markers of inflammation, and cellular aging in older adult AD spousal caregivers with insomnia (N=150) over one-year follow-up. The specific aims of this project are:

Primary Aim 1: Determine the effects of MAP-I vs. CBT-I on subjective and objective dimensions of insomnia.

Secondary Aim 1: Evaluate the effects of MAP-I vs. CBT-I on cellular and genomic markers of inflammation.

Secondary Aim 2: Evaluate the effects of MAP-I vs. CBT-I on markers of cellular aging.

Exploratory Aim 1: Explore moderating effects of caregiver stress (Stress and Adversity Inventory, STRAIN, number & experienced intensity of stress exposure) on insomnia outcomes, and effects of MAP-I vs. CBT-I on caregiver stress, health functioning, chronic medical morbidity and related medication use at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer or other dementia caregivers
* Older than 45 years of age
* Self-identified as the principal person taking care of the patient with Alzheimer or other dementia
* Diagnostic and Statistical Manual Criteria - 5 for Insomnia

Exclusion Criteria:

* Psychiatric disorders including current major depressive disorder or other current DSM-5 psychiatric disorder (e.g. substance dependence) with the exception of anxiety disorder;
* Psychotic symptoms;
* Acute suicidal or violent behavior or history of suicide attempt within the last year
* Other sleep disorders including current or lifetime history of sleep apnea, nocturnal myoclonus, phase-shift disorder as identified by SCID-5 and Duke Structured Interview for Sleep Disorders (DSISD)
* Medical conditions such as acute or uncontrolled medical illness (e.g., major surgery, metastatic cancer, Class III heart failure, inflammatory disorder)
* Chronic infections
* Obesity with body mass index (BMI) >35
* Use of hormone containing medications including steroids or immune modifying drugs
* Daily use of analgesics such as opioids;
* Daily us of sedative hypnotic medications
* Cognitive impairment as evidenced by DSM-5 interview and/or Mini-Mental Status Exam (MMSE < 26)
* Actively practicing a mind body intervention.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Insomnia clinical response | One-year
  Change in severity of insomnia as measured by the Insomnia Severity Index

SECONDARY OUTCOMES:
Insomnia clinical response | One year
  Change in severity of insomnia as measured by clinical diagnosis
Daytime dysfunction | One year
  Change in depressed mood as measured by the Inventory of Depressive Symptoms
Inflammation | One year
  Change in markers of systemic inflammation as measured by C-reactive protein
Cellular aging | One year
  Change in markers of cellular aging as measured by transcriptional profiles of the senescent secretory associated phenotype (SASP)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Irwin, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided